CLINICAL TRIAL: NCT04564625
Title: Relationships Between Vitamin D and Orthopedic Trauma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 005.TRA.2020.D
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Fracture; Fracture Nonunion; Fractures, Bone; Vitamin D
Keywords: fracture; fracture nonunion; vitamin D
MeSH Terms: conditions — Fractures, Bone; Fractures, Ununited

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fracture and Vitamin D assessment: All patients between 18 and 25 years treated for fractures at Methodist Dallas Medical Center (MDMC) with an index admission vitamin D assessment will be enrolled. This study will consider any patients with an index admission occurring between February 2016 and February 2020. No changes to care or intervention will occur and this study will be conducted completely via chart review. The aim is to identify 100 subjects with a one-year follow-up appointment for their injury to determine the rate of nonunion and vitamin D levels. As patients receive vitamin D supplementation as standard of care if index values are low, impact will be assessed through relative deficiency and clinical outcomes. Data collected from subjects without need for supplementation may be used to generate a threshold.
  Interventions: Other: Vitamin D Assessment; Other: Fracture

INTERVENTIONS:
Other: Vitamin D Assessment — index admission vitamin D assessment
Other: Fracture — rate of nonunion (i.e., failure of a fractured bone to heal)

SUMMARY:
Vitamin D is an essential hormone involved in bone metabolism, bone mineral density maintenance, and bone health. Vitamin D deficiency is putatively linked to poor pediatric orthopedic outcomes [1]. Further, the risk of low vitamin D associated fractures may be greater in minority pediatric populations [2]. In adults, utility of vitamin D alleles as a biomarker for bone density and fracture risk has been debated for over 10 years [3-5]. Peak bone density is achieved at 25 years old; however, most orthopedic trauma patients less than 25 years of age present with substantial vitamin D deficiencies.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1. Background Vitamin D is an essential hormone involved in bone metabolism, bone mineral density maintenance, and bone health. Vitamin D deficiency is putatively linked to poor pediatric orthopedic outcomes [1]. Further, the risk of low vitamin D associated fractures may be greater in minority pediatric populations [2]. In adults, utility of vitamin D alleles as a biomarker for bone density and fracture risk has been debated for over 10 years [3-5]. Peak bone density is achieved at 25 years old; however, most orthopedic trauma patients less than 25 years of age present with substantial vitamin D deficiencies.

   1.2. Aim(s)
   * Identify the prevalence of vitamin D deficiency in young trauma patients with fractures.
   * Describe the merits of vitamin D supplementation in healing and long-term outcomes ≤25 year old trauma patients with fractures.

   1.3. Rationale for the study Occurrence of stress and low energy mechanism fractures within a population at peak bone density is troubling and suggestive of underlying pathology. Understanding how to combat vitamin D deficiency, and improve outcomes, is essential in the development of comprehensive and preventative trauma care.

   1.4. Hypothesis 1.4.1. Primary Hypothesis Patients aged ≤25yrs old with fractures will have low vitamin-D levels.
2. OBJECTIVES AND STUDY OUTCOME MEASURES 2.1. Study Objectives 2.1.1. Primary Objective Determine the frequency of vitamin D deficiency in fracture patients aged less than 25 years old.

   2.1.2. Secondary Objective Report the long-term (one year) outcomes for fracture healing relative to baseline and therapeutic vitamin D levels.

   2.2. Study Outcome Measures 2.2.1. Primary Outcome Vitamin D levels at the time of the index injury through one year post-operative follow up.

   2.2.2. Secondary Outcomes Patient demographics (age, sex, ethnicity), injury characteristics, lab values, rate of nonunion (i.e., failure of a fractured bone to heal), admit information, discharge disposition, payer type, and mortality.
3. STUDY DESIGN All patients between 18 and 25 years treated for fractures at Methodist Dallas Medical Center (MDMC) with an index admission vitamin D assessment will be enrolled. This study will consider any patients with an index admission occurring between February 2016 and February 2020. No changes to care or intervention will occur and this study will be conducted completely via chart review. The aim is to identify 100 subjects with a one-year follow-up appointment for their injury to determine the rate of nonunion and vitamin D levels. As patients receive vitamin D supplementation as standard of care if index values are low, impact will be assessed through relative deficiency and clinical outcomes. Data collected from subjects without need for supplementation may be used to generate a threshold. Patient demographics will be considered as practice suggests minority patients may be disproportionally affected. The plan to complete the data collection and analysis by February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >18 years old and ≤25 years old
* Patients must have any fracture requiring follow-up
* Patients must have received vitamin-D assessment

Exclusion Criteria:

* Patients aged >25yrs
* Prisoners
* Pregnant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients between 18 and 25 years treated for fractures at Methodist Dallas Medical Center (MDMC) with an index admission vitamin D assessment will be enrolled. This study will consider any patients with an index admission occurring between February 2016 and February 2020.We will also consider patient demographics as practice suggests minority patients may be disproportionally affected.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels at the time of the index injury through one year post-operative follow up. | February 2016 and February 2020
  Vitamin D levels at the time of the index injury through one year post-operative follow up.

SECONDARY OUTCOMES:
Patient demographics | February 2016 and February 2020
  age, sex, ethnicity
injury characteristics | February 2016 and February 2020
  injury characteristics
rate of nonunion | February 2016 and February 2020
  failure of a fractured bone to heal
admit information | February 2016 and February 2020
  admit information
discharge disposition | February 2016 and February 2020
  discharge disposition
payer type | February 2016 and February 2020
  payer type
mortality | February 2016 and February 2020
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Araiza, MD, Principal Investigator — Methodist
Locations (1):
- Methodist Health System Clinical Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a single center study and the data will not be shared with outside entities until it is de-identified in order to be presented at relevant conferences or published in a scientific journal

REFERENCES:
- [Background] Horan MP, Williams K, Hughes D. The Role of Vitamin D in Pediatric Orthopedics. Orthop Clin North Am. 2019 Apr;50(2):181-191. doi: 10.1016/j.ocl.2018.10.002. PMID 30850077
- [Background] Ramirez N, Ortiz-Fullana JL, Arciniegas N, Fullana A, Valentin P, Orengo JC, Iriarte I, Carlo S. Vitamin D levels and fracture risk among Hispanic children. Eur J Orthop Surg Traumatol. 2019 Apr;29(3):531-536. doi: 10.1007/s00590-018-2315-7. Epub 2018 Oct 13. PMID 30317468
- [Background] McClean E, Archbold GP, Taggart HM. Do the COL1A1 and Taq 1 vitamin D receptor polymorphisms have a role in identifying individuals at risk of developing osteoporosis? Ulster Med J. 2003 May;72(1):26-33. PMID 12868700
- [Background] Lorentzon M, Lorentzon R, Nordstrom P. Vitamin D receptor gene polymorphism is associated with birth height, growth to adolescence, and adult stature in healthy caucasian men: a cross-sectional and longitudinal study. J Clin Endocrinol Metab. 2000 Apr;85(4):1666-70. doi: 10.1210/jcem.85.4.6566. PMID 10770213
- [Background] Ensrud KE, Stone K, Cauley JA, White C, Zmuda JM, Nguyen TV, Eisman JA, Cummings SR. Vitamin D receptor gene polymorphisms and the risk of fractures in older women. For the Study of Osteoporotic Fractures Research Group. J Bone Miner Res. 1999 Oct;14(10):1637-45. doi: 10.1359/jbmr.1999.14.10.1637. PMID 10491209